CLINICAL TRIAL: NCT00590902
Title: Multicenter Phase II Trial of OSI-774 (Erlotinib, Tarceva) In Patients With Advanced Bronchioloalveolar Cell Lung Cancer
Brief Title: Ph II OSI-774 (Erlotinib,Tarceva) In Advanced Bronchioloalveolar Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Northwestern University (Other); Vanderbilt-Ingram Cancer Center (Other); Dana-Farber Cancer Institute (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-010
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Bronchioloalveolar Cell Variant of Non-small Cell Lung Cancer
Keywords: non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 - OSI-774 (Experimental)
  Interventions: Drug: OSI-774: erlotinib, TarcevaTM

INTERVENTIONS:
Drug: OSI-774: erlotinib, TarcevaTM — 150 mg, 100 mg and 25 mg tablets

SUMMARY:
The primary objective of this study is to determine the major objective response rate of OSI-774 in participants with unresectable or metastatic bronchioloalveolar cell variant of non-small cell lung cancer.

This study is a Phase II study. The first study of OSI-774 was done to evaluate what dose should be given to patients with cancer has been completed. The purpose of this research study is to see whether this experimental treatment, called OSI-774, can cause a type of non-small cell lung cancer to stop growing or shrink. This study is sponsored by a company called Genentech, and is being done at Memorial Hospital, as well as other cancer centers around the country interested in developing new drugs for the treatment of this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Either bronchioloalveolar cell carcinoma or a variant thereof after review
* Clinical stage IIIB (malignant pleural or pericardial effusion) or IV or recurrent/medically inoperable disease
* Measurable or evaluable indicator lesions
* No prior or one chemotherapy regimen for NSCLC
* Three weeks since last chemotherapy, and three weeks since prior radiation therapy to a major bone-marrow containing area
* Karnofsky performance status > or = to 80% OR ECOG performance status ≤ or = to 1
* Life expectancy > or = to 8 weeks
* Adequate hematologic, renal and/or hepatic function: WBC > or = to 3,000/ul, hemoglobin > or = to 9.0 g/dl, platelet count > or = to 100,000/ul, total bilirubin < or = to 1.0 mg/dl, AST < than or = to 2.5 X UNL, creatinine < or = to 1.5 mg/dl or Clcr > or = to 55ml/min.
* Effective contraception

Exclusion Criteria:

* Prior exposure to OSI-774 or other treatments targeting the HER family axis (e.g.-trastuzumab, ZD1839, C225, etc.)
* Two or more prior chemotherapy regimens
* Concurrent active cancer
* Uncontrolled central nervous system metastases (i.e. any known CNS lesion which is radiographically unstable, symptomatic and/or requiring escalating doses of corticosteroids)
* Pregnant or lactating women
* Malignancies within the past 5 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Prior systemic cytotoxic chemotherapy for other malignant disease
* Significant medical history or unstable medical condition (unstable systemic disease: congestive heart failure, recent MI, unstable angina, active infection, uncontrolled hypertension).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2002-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Azzoli, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 - OSI-774
Started | 81
Completed | 80
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1 - OSI-774
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response of OSI-774
Description: (complete and partial responses) Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. A complete response is the disappearance of all target lesions, and a partial response (PR) is defined as at least a 30% decrease in the sum of the target lesions. Stable disease is defined as fitting the criteria neither for progressive disease nor a PR.
Time Frame: 53 weeks
Measure: Number; unit: participants
Arm/Group | 1 - OSI-774
Number analyzed (Participants) | 80
participants
  Complete Response (CR) | 1
  Partial Response (PR) | 18
  Stable Disease (SD) | 31
  Progression of Disease (POD) | 30

ADVERSE EVENTS:
Arm/Group | 1 - OSI-774
Serious Adverse Events (participants affected / at risk) | 22/81
Other Adverse Events (participants affected / at risk) | 66/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - OSI-774 (N=81)
Abdominal pain/cramping (Gastrointestinal disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Headache (General disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Mood alteration - Agitation (Nervous system disorders) | 1 (1)
Mood alteration - Anxiety (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neurology, other (Nervous system disorders) | 1 (1)
Neuropathy-sensory (Nervous system disorders) | 1 (1)
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vision-double vision (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - OSI-774 (N=81)
Bilirubin (Metabolism and nutrition disorders) | 22 (22)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (17)
Dermatology, skin other (Skin and subcutaneous tissue disorders) | 10 (16)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (24)
Fatigue (General disorders) | 20 (22)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 5 (5)
Rash, desquamation (Skin and subcutaneous tissue disorders) | 28 (44)
SGPT (ALT) (Blood and lymphatic system disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes